CLINICAL TRIAL: NCT07347171
Title: A Phase 1, Open-label, Multicentre Study Evaluating the Safety, Tolerability, Pharmacokinetic/Pharmacodynamic Characteristics, and Preliminary Efficacy of CG009301 for Injection in Adult Subjects With Relapsed or Refractory Haematological Malignancies
Brief Title: A Phase 1 Study of CG009301 for Injection in Adult Subjects With Recurrent or Refractory Haematological Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cullgen (Shanghai),Inc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG-GSPT1-9301001; CTR20244643 (Other: ChinaDrugTrials)
Record Dates: First submitted 2025-12-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Leukemia; AML; MDS; AML (Acute Myelogenous Leukemia); MDS (Myelodysplastic Syndrome)
Keywords: Leukemia; GSPT1; CG009301; AML; MDS
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- 0.25mg QD (Experimental): CG009301 for Injection
  Interventions: Drug: CG009301 for Injection
- 0.5mg QD (Experimental): CG009301 for Injection
  Interventions: Drug: CG009301 for Injection
- 1.0mg QD (Experimental): CG009301 for Injection
  Interventions: Drug: CG009301 for Injection
- 1.6mg QD (Experimental): CG009301 for Injection
  Interventions: Drug: CG009301 for Injection
- 2.5mg QD (Experimental): CG009301 for Injection
  Interventions: Drug: CG009301 for Injection
- 3.5mg QD (Experimental): CG009301 for Injection
  Interventions: Drug: CG009301 for Injection
- 5.0mg QD (Experimental): CG009301 for Injection
  Interventions: Drug: CG009301 for Injection
- 6.5mg QD (Experimental): CG009301 for Injection
  Interventions: Drug: CG009301 for Injection
- 8.25mg QD (Experimental): CG009301 for Injection
  Interventions: Drug: CG009301 for Injection
- 10.0mg QD (Experimental): CG009301 for Injection
  Interventions: Drug: CG009301 for Injection

INTERVENTIONS:
Drug: CG009301 for Injection — 0.9% Sodium Chloride Injection diluted to 250mL，Cycle 1 and subsequent cycles, IV, infusion duration: 2 hours, once daily (QD) administration for 7 days continuously(28 days constituting one cycle)

SUMMARY:
The goal of this clinical trial is to learn about the safety of drug CG009301. It also learns if drug CG009301 works to treat in Participants with relapsed or refractory adult haematological malignancies.

The main question[s] it aims to answer are:

1. To determine the maximum tolerated dose (MTD) and/or objective best dose (OBD) of CG009301 for injection in subjects with relapsed or refractory adult haematological malignancies.
2. To establish subsequent dosing regimens for CG009301 for injection.
3. To characterise the safety profile and tolerability of CG009301 for injection. Participants will Receive treatment with CG009301 until disease progression.

DETAILED DESCRIPTION:
This study will employ a multicentre, open-label design to evaluate the safety, tolerability, pharmacokinetic/pharmacodynamic characteristics, and preliminary efficacy of CG009301 for injection in adult subjects with relapsed or refractory haematological malignancies.

This Phase I trial will comprise two phases, corresponding to the following indications:

Dose-escalation study - Relapsed/refractory haematological malignancies, regardless of tumour type; Dose-expansion phase: Relapsed/refractory (R/R) acute myeloid leukaemia (AML), high-risk myelodysplastic syndromes (HR-MDS), and R/R acute lymphoblastic leukaemia (ALL).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and <75 years at the time of signing the informed consent form; no gender restrictions;
2. Patients with relapsed/refractory haematological malignancies who have received a definitive diagnosis by pathology and/or cytology, confirmed histologically, and who have failed prior standard treatment regimens. The investigator must deem that no standard treatment is available or that the patient cannot tolerate existing therapies. Dose-escalation phase: unrestricted haematological tumour types. Dose-expansion phase: must meet one of the following criteria: a. Subjects meeting AML diagnostic criteria based on WHO 2022 5th edition classification, confirmed by bone marrow cytomorphology, including AML evolving from early-stage MDS or MPN. Criteria for recurrent AML: Leukaemic cells reappearing in peripheral blood after CR, or >5% blast/immature cells in bone marrow, or extramedullary leukaemic infiltration. Criteria for refractory AML: - Treatment-naïve cases unresponsive to two standard-regimen cycles; - Relapse within 12 months after consolidation/intensification therapy following CR; - Relapse after 12 months unresponsive to conventional chemotherapy; Patients with two or more relapses; Persistent extramedullary leukaemia; b. Patients diagnosed with high-risk or very high-risk MDS according to the WHO 2022 5th edition classification, with a percentage of blasts in bone marrow smear or biopsy pathology < 20%, and deemed by the investigator to have no other appropriate treatment options. Diagnostic criteria for recurrent MDS: Following achievement of complete remission, partial remission, or haematological improvement, at least one of the following must occur: - Bone marrow blastic count returns to pre-treatment levels; - ANC or PLT decreases by ≥50% from best response; - HGB decreases by ≥15 g/L or becomes transfusion-dependent. Diagnostic criteria for refractory MDS: Following adequate treatment (at least four cycles of demethylating agent therapy), meeting the IWG 2023 response criteria for "stable disease", "failure", or "disease progression"; progression after demethylating agent or other drug therapy, or patient intolerance to toxicity (e.g., treatment-related grade 3 or higher hepatic or renal toxicity during therapy leading to permanent discontinuation); c. Subjects meeting ALL diagnostic criteria based on WHO 2022 5th edition classification, with ≥20% primitive/immature lymphocytes in bone marrow. Relapsed ALL diagnostic criteria: Patients who, after achieving CR following induction therapy, exhibit recurrence of leukaemic cells in peripheral blood, >5% primitive/immature lymphocytes in bone marrow, or development of extramedullary disease; Criteria for refractory ALL: Patients failing to achieve CR following standard induction therapy;
3. ECOG performance status score of 0-1;
4. Investigator-assessed expected survival ≥3 months;
5. Recovery of toxicities from prior treatment to ≤Grade 1 according to NCI-CTCAE v5.0 (excluding alopecia and long-term stable chronic conditions);
6. No prior autologous haematopoietic stem cell transplantation, or transplantation more than 2 months prior with toxicities resolved to ≤ Grade 1;
7. Adequate organ function support, with screening laboratory tests meeting all criteria: a. Coagulation function prior to study drug administration: INR ≤ 1.5 × ULN or aPTT ≤ 1.5 × ULN; b. Hepatic function: serum total bilirubin ≤ 2× ULN; AST and/or ALT ≤ 2.5× ULN; c. Cr ≤ 2× ULN or CrCL > 30 mL/min (calculated using Cockcroft-Gault formula); d. LVEF ≥ 40%; and QTc ≤ 480 milliseconds; e. White blood cell count may decrease below 50.0 × 10⁹/L at baseline or following hydroxyurea administration
8. Non-pregnant and non-lactating: Infertile subjects; or subjects with potential for conception who agree to use effective contraception (hormonal, barrier, or abstinence). Male subjects must also abstain from sperm donation during study participation and for 90 days after the last dose of CG009301 injection. Women of childbearing potential must have a negative serum pregnancy test (serum-β-hCG) during the screening period;
9. Understand the study's purpose, process, nature, significance, potential benefits, and risks, and voluntarily sign the written informed consent form. Be able to comply with scheduled visits, treatment plans, laboratory tests, and other study instructions or procedures.

Exclusion Criteria:

1. Central nervous system leukaemia presenting with neurological and/or psychiatric symptoms;
2. Receipt of antitumour therapy (excluding hydroxyurea and prophylactic intrathecal injections) such as chemotherapy, immunotherapy, targeted therapy, or biological therapy within 4 weeks or 5 half-lives (whichever is shorter) prior to the first study drug administration; receipt of radiotherapy within 2 weeks; receipt of traditional Chinese herbal medicine within 2 weeks;
3. Major surgery within 4 weeks prior to the first study dose, or anticipated need for major surgery during the study period;
4. Active infection deemed uncontrolled by the investigator following treatment with antibiotics, antiviral agents, or antifungal medications;
5. Severe or uncontrolled underlying medical conditions deemed ineligible for inclusion by the investigator, including but not limited to respiratory disorders (e.g., chronic obstructive pulmonary disease requiring oxygen therapy, moderate or higher asthma, moderate or higher pulmonary fibrosis, recurrent pulmonary oedema), cardiovascular disorders (e.g., prior coronary artery bypass grafting or coronary stent implantation, myocardial infarction within the past 6 months, NYHA Class III-IV heart failure), unstable angina within the past 6 months, uncontrolled hypertension (systolic >160 mmHg or diastolic >100 mmHg), arrhythmias requiring ongoing medical or interventional management), endocrine disorders (severe hyperthyroidism/hypothyroidism, uncontrolled diabetes mellitus), and neurological/psychiatric conditions affecting cognition, compliance, or personal safety (e.g., unstable epilepsy, dementia, schizophrenia, depression); psychiatric disorders (e.g., unstable epilepsy, dementia, schizophrenia, depression);
6. Active autoimmune diseases (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune haemolytic anaemia, scleroderma, severe psoriasis, rheumatoid arthritis), or allergy to the study drug or excipients;
7. Significant non-leukaemia-related bleeding risk (e.g., anticoagulant or antiplatelet therapy, arteriovenous malformation), or recent history of major bleeding (e.g., gastrointestinal haemorrhage, intracranial haemorrhage, disseminated intravascular coagulation);
8. Grade 2 or higher central nervous system or peripheral neuropathy (excluding stable Grade 3 conditions lasting over 6 months that do not impair daily functioning);
9. Allogeneic haematopoietic stem cell transplantation within 12 months prior to initial administration;
10. History of deep vein thrombosis, pulmonary embolism, or any other severe thromboembolic event within 6 months prior to initial administration (thrombosis originating from implanted venous access ports or catheters, superficial vein thrombosis, or lacunar cerebral infarction are not considered "severe" thromboembolic events); Known familial and/or acquired thrombotic predisposition, such as hereditary or acquired defects in anticoagulant proteins, coagulation factors, fibrinolytic proteins, or presence of acquired risk factors conferring high thrombotic propensity;
11. HIV, HBV, and HCV infection: positive HIV antibody and PCR tests; HBsAg positive or viral DNA ≥100 IU/mL; positive HCV antibody with HCV-RNA quantification exceeding the upper limit of normal;
12. Individuals who received (attenuated) live virus vaccination within 4 weeks prior to first dosing;
13. Individuals with a documented history of alcohol or substance abuse;
14. Any past or current medical condition, treatment, or laboratory abnormality that may interfere with study results or affect the subject's ability to complete the study, or if the investigator deems the subject unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The RDE(Recommended Dose for Expansion)of CG009301 for injection. | up to 8 months
  RDE refer to recommended dose for expansion
Duration of continuous administration and dosing cycle for CG009301 for injection | up to 20 months
Safety profile of CG009301 for injection: Incidence, severity, duration, outcome, and relationship to the study drug for adverse events (AEs), serious adverse events (SAEs), dose-limiting toxicity (DLT), and clinically significant laboratory abnormalitie | up to 20 months

SECONDARY OUTCOMES:
Cmax | up to 20 months
  Cmax refer to Peak concentration
Tmax | up to 20 months
  Tmax refer to Time to peak concentration
AUC0-t | up to 20 months
  AUC0-t refer to Area under the concentration-time curve from zero to the last quantifiable time point
AUCinf | up to 20 months
  AUCinf refer to Area under the concentration-time curve from zero extrapolated to infinity
T1/2 | up to 20 months
  T1/2 refer to Half-life
CL | up to 20 months
  CL refer to Apparent clearance
Vd | up to 20 months
  Vd refer to Apparent volume of distribution
Cmax,ss | up to 20 months
  Cmax,ss refer to Steady-state peak concentration
Cmin,ss | up to 20 months
  Cmin,ss refer to Steady-state trough concentration
drug accumulation ratio | up to 20 months
ORR | up to 20 months
  ORR refer to objective response rate, the proportion of subjects whose best overall response is CR(complete response),CRi(complete response with incomplete hematologic recovery),CRh(complete remission with partial hematologic recovery), MLFS(morphologic leukemia-free state) or PR(partial response) in the study assessed by investigator according to response criteria of hematological malignancy,which AML(Acute Myeloid Leukemia) according to 2022 European LeukemiaNet (ELN) Response Criteria for Acute Myeloid Leukemia(Döhner et al., Blood 2022),ALL(Acute Lymphoblastic Leukemia) according to National Comprehensive Cancer Network. NCCN Clinical Practice Guidelines in Oncology: Acute Lymphoblastic Leukemia(Version 4.2023).,MDS(Myelodysplastic Syndromes) according to International Working Group 2023 response criteria for higher-risk myelodysplastic syndromes(Zeidan AM et al., Blood 2023).
CRR | up to 20 months
  CRR refer to complete response rate, the proportion of subjects whose best overall response is CR(complete response),CRi(complete response with incomplete hematologic recovery) or CRh(complete remission with partial hematologic recovery)in the study assessed by investigator according to response criteria of hematological malignancy,which AML(Acute Myeloid Leukemia) according to 2022 European LeukemiaNet (ELN) Response Criteria for Acute Myeloid Leukemia(Döhner et al., Blood 2022),ALL(Acute Lymphoblastic Leukemia) according to National Comprehensive Cancer Network. NCCN Clinical Practice Guidelines in Oncology: Acute Lymphoblastic Leukemia(Version 4.2023).,MDS(Myelodysplastic Syndromes) according to International Working Group 2023 response criteria for higher-risk myelodysplastic syndromes(Zeidan AM et al., Blood 2023).
EFS | up to 92 months
  EFS refer to Event-Free Survival. Defined as the time from the first administration of CG009301 to the first occurrence of trail failure,disease relapse after CR(complete response),CRi(complete response with incomplete hematologic recovery) or CRh(complete remission with partial hematologic recovery), or death (whichever occurs first), as assessed by the investigator according to response criteria of hematological malignancy,which AML according to 2022 European LeukemiaNet (ELN) Response Criteria for Acute Myeloid Leukemia(Döhner et al., Blood 2022),ALL according to National Comprehensive Cancer Network. NCCN Clinical Practice Guidelines in Oncology: Acute Lymphoblastic Leukemia(Version 4.2023).,MDSaccording to International Working Group 2023 response criteria for higher-risk myelodysplastic syndromes(Zeidan AM et al., Blood 2023).
  Trail failure defined as didn't achieve CR,CRi or CRh after 6 period treatment.
RFS | up to 92 months
  RFS refer to Relapse-Free Survival. Only uesd to evaluate the subjects which achieved CR(complete response),CRi(complete response with incomplete hematologic recovery) or CRh(complete remission with partial hematologic recovery),Defined as the time from the day subject achieve CR,CRi or CRh,to the hematologic relapse or death (whichever occurs first),as assessed by the investigator according to response criteria of hematological malignancy,which AML according to 2022 European LeukemiaNet (ELN) Response Criteria for Acute Myeloid Leukemia(Döhner et al., Blood 2022),ALL according to National Comprehensive Cancer Network. NCCN Clinical Practice Guidelines in Oncology: Acute Lymphoblastic Leukemia(Version 4.2023).,MDSaccording to International Working Group 2023 response criteria for higher-risk myelodysplastic syndromes(Zeidan AM et al., Blood 2023).
Determination of the RP2D for CG009301 for Injection | up to 20 months
  RP2D refer to recommended phase 2 dose

OTHER OUTCOMES:
Pharmacodynamics: Degree of GSPT1 protein degradation in peripheral blood mononuclear cells following administration of injectable CG009301 at different doses. | up to 20 months
CCR MRD negative | up to 20 months
  MRD refer to minimal residual disease,which can be tested by flow cytometry. CCR MRD negative defined as among the subjects achieved CR(complete response),CRi(complete response with incomplete hematologic recovery) or CRh(complete remission with partial hematologic recovery),the rate of the subjects achieved MRD negative.
EFS MRD negative | up to 92 months
  MRD refer to minimal residual disease,which can be tested by flow cytometry.Only uesd for the subjects achieved CR(complete response),CRi(complete response with incomplete hematologic recovery) or CRh(complete remission with partial hematologic recovery), and the subjects achieved MRD negative.Defined as the time from the first administration of CG009301 to the first occurrence of trail failure,hematologic relapse or extramedullary relapse,MRD relapse or death (whichever occurs first), as assessed by the investigator according to response criteria of hematological malignancy.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, MS, Principal Investigator — The Haematology Hospital of the Chinese Academy of Medical Sciences
Locations (3):
- China (3):
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Haematology Hospital of the Chinese Academy of Medical Sciences, Tianjin
  - Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: No